CLINICAL TRIAL: NCT05260021
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study With an Open-Label Extension Assessing the Efficacy, Safety, and Pharmacokinetics/Pharmacodynamics of Tirzepatide in Pediatric and Adolescent Participants With Type 2 Diabetes Mellitus Inadequately Controlled With Metformin, or Basal Insulin, or Both
Brief Title: A Study to Evaluate Tirzepatide (LY3298176) in Pediatric and Adolescent Participants With Type 2 Diabetes Mellitus Inadequately Controlled With Metformin or Basal Insulin or Both
Acronym: SURPASS-PEDS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17121; I8F-MC-GPGV (Other: Eli Lilly and Company); 2021-003612-31 (EudraCT Number)
Record Dates: First submitted 2022-02-25; First posted 2022-03-02 (Actual); Results first posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Type2 Diabetes; Diabetes Mellitus; Diabetes Mellitus, Type 2; T2D; T2DM (Type 2 Diabetes Mellitus); Glucose Metabolism Disorders; Endocrine System Diseases; Metabolic Disease
Keywords: GLP-1 RA; Glucose-dependent insulinotropic polypeptide (GIP); glucagon-like peptide-1 (GLP-1); GIP/GLP-1 dual receptor agonist; Incretins
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Endocrine System Diseases; Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tirzepatide Dose 1 (Experimental): Double-Blind:
  Participants receive Tirzepatide by weekly subcutaneous (SC) injection starting with a low dose then increase to a higher dose every four weeks until maintenance dose level 1 is reached.
  Open-Label:
  Participants will continue to receive Tirzepatide at the last dose level
  Interventions: Drug: Tirzepatide Dose 1
- Tirzepatide Dose 2 (Experimental): Double-Blind:
  Participants receive Tirzepatide by weekly SC injection starting with a low dose then increase to a higher dose every four weeks until maintenance dose level 2 is reached.
  Open-Label:
  Participants will continue to receive Tirzepatide at the last dose level
  Interventions: Drug: Tirzepatide Dose 2
- Placebo (Placebo Comparator): Double-Blind:
  Participants receive placebo during the 30-week double-blind period.
  Open-Label:
  Participants will switch to Tirzepatide by weekly SC injection starting with a low dose then increase to a higher dose every four weeks until maintenance dose level 1 is reached.
  Interventions: Drug: Tirzepatide Dose 1; Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide Dose 1 — Administered SC
  Arms: Placebo; Tirzepatide Dose 1
Drug: Tirzepatide Dose 2 — Administered SC
  Arms: Tirzepatide Dose 2
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn more about the safety and efficacy of tirzepatide compared to placebo in children or teenagers with type 2 diabetes taking metformin, or basal insulin, or both.

The overall study will last about 60 weeks with up to 14 clinic visits and 6 phone visits. Clinic visits will include blood sample collection, physical exam and questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 10 to below 18 years at screening visit
* Have type 2 diabetes, treated with diet and exercise and metformin and/or basal insulin. Metformin and/or basal insulin dose must be stable for at least 90 days prior to study screening.
* Have HbA1c >6.5% to ≤11% at screening
* Have body weight ≥50 kilogram (kg) 110 pounds and BMI of >85th percentile of the general age and gender-matched population for that country or region.

Exclusion Criteria:

* Have Type 1 diabetes mellitus (T1DM), or positive GAD65 or IA2 antibodies
* After the T2DM diagnosis, have a history of diabetic ketoacidosis or hyperosmolar syndrome
* Have had ≥1 episode of severe hypoglycemia and/or ≥1 episode of hypoglycemic unawareness within the last 6 months.
* Have family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN2).
* Had chronic or acute pancreatitis any time prior to study entry
* Female participants who are pregnant or breast feeding or intending to become pregnant.
* Using prescription or over the counter medications for weight loss within 90 days of the screening visit.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 99 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2025-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: 1-877-CTLilly (1877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (51):
- United States (13):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Center Of Excellence in Diabetes and Endocrinology, Sacramento, California
  - Rady Children's Hospital, San Diego, California
  - Touro University California, Vallejo, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Children's Health - Delaware, Wilmington, Delaware
  - Qualmedica Research, LLC, Evansville, Indiana
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - AA Medical Research Center, Flint, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - SUNY Upstate Medical University, Syracuse, New York
  - Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - Consano Clinical Research, LLC, Shavano Park, Texas
- Australia (3):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Centre for Children's Health Research, Brisbane, Queensland
  - Perth Children's Hospital, Perth, Western Australia
- Brazil (11):
  - CEDOES, Vitória, Espírito Santo
  - Centro de Diabetes Curitiba, Curitiba, Paraná
  - Instituto Méderi de Pesquisa e Saúde, Passo Fundo, Rio Grande do Sul
  - Instituto da Crianca com Diabetes, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa Sao Lucas, Campinas, São Paulo
  - Instituto de Pesquisa clinica de Campinas, Campinas, São Paulo
  - Instituto de Pesquisa Clinica, São Paulo, São Paulo
  - Instituto da Crianca do Hospital das Clinicas da FMUSP, São Paulo, São Paulo
  - Ruschel Medicina e Pesquisa Clínica, Rio de Janeiro
  - CPQuali Pesquisa Clínica, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
- France (2):
  - Centre Hospitalier Universitaire d'Angers, Angers, Maine-et-Loire
  - Assistance Publique - Hopitaux de Paris (AP-HP) - Hopital Robert Debre - Centre Hospitalo Universitaire (C -T, Paris
- India (6):
  - Gujarat Endocrin Pvt Ltd, Ahmedabad, Gujarat
  - M S Ramaiah Medical College and Hospitals, Bangalore, Karnataka
  - Bhakti Vedanta Hospital and Research Institute, Thane, Maharashtra
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Kovai Diabetes Speciality Center and Hospital, Coimbatore, Tamil Nadu
  - Postgraduate Institute of Medical Education & Research, Chandigarh
- Israel (5):
  - Yitzhak Shamir Medical Center, Be’er Ya‘aqov, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Shaare Zedek Medical Center, Jerusalem, Jerusalem
  - Rambam Health Care Campus, Haifa, Northern District
  - Soroka Medical Center, Beersheba, Southern District
- Italy (3):
  - Azienda Ospedaliera Universitaria dell'Università "Luigi Vanvitelli" Piazza Luigi Miraglia, 2 Napoli Campa -T, Napoli, Campania
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Trento, Verona, Veneto
  - Ospedale Pediatrico Salesi, Ancona
- Mexico (5):
  - Unidad Médica para la Salud Integral, San Nicolás de los Garza, Nuevo León
  - Clínica Cemain, Tampico, Tamaulipas
  - Investigacion En Salud Y Metabolismo Sc, Chihuahua City
  - Consultorio Médico de Endocrinología y Pediatría, Puebla City
  - Arké SMO S.A de C.V, Veracruz
- United Kingdom (3):
  - Leicester Royal Infirmary, Leicester, England
  - Hull Royal Infirmary, Hull, Kingston Upon Hull
  - Leicester General Hospital, Leicester, Leicestershire

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Hannon TS, Chao LC, Barrientos-Perez M, Pamidipati KC, Lando LF, Lee CJ, Patel H, Bergman BK. Efficacy and safety of tirzepatide in children and adolescents with type 2 diabetes (SURPASS-PEDS): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2025 Oct 4;406(10511):1484-1496. doi: 10.1016/S0140-6736(25)01774-X. Epub 2025 Sep 17. PMID 40975112
- See also: A Study to Evaluate Tirzepatide (LY3298176) in Pediatric and Adolescent Participants With Type 2 Diabetes Mellitus Inadequately Controlled With Metformin or Basal Insulin or Both (SURPASS-PEDS) — https://trials.lillytrialguide.com/en-US/trial/WoqX8k1IVNPugq1V1yyyL

RESULTS

PARTICIPANT FLOW:
Groups:
- 5 Milligram (mg) Tirzepatide/5 mg Tirzepatide: Participants received 5 mg Tirzepatide once weekly (QW) administered as subcutaneous (SC) injection via single-dose pen (SDP) for 30 weeks in double-blind period and 22 weeks in open-label period with an additional 4 weeks of safety follow-up.
- 10 mg Tirzepatide/10 mg Tirzepatide: Participants received 10 mg Tirzepatide QW administered as SC injection via SDP for 30 weeks in double-blind period and 22 weeks in open-label period with an additional 4 weeks of safety follow-up.
- Placebo/5 mg Tirzepatide: Participants received placebo QW administered as SC injection via SDP for 30 weeks in double-blind period and 5 mg Tirzepatide QW administered as SC injection via SDP for 22 weeks in open-label period.
Period: Double-blind Period (30 Weeks)
Arm/Group | 5 Milligram (mg) Tirzepatide/5 mg Tirzepatide | 10 mg Tirzepatide/10 mg Tirzepatide | Placebo/5 mg Tirzepatide
Started | 32 | 33 | 34
Received Atleast One Dose of Study Drug | 32 | 33 | 34
Safety Analysis Set 1 (Safety Analysis set 1 is defined as, data obtained from mITT participants (those who took at least 1 dose of study intervention was included in the analyses) during Double blind period, regardless of adherence to study intervention or initiation of rescue antihyperglycemic medication.) | 32 | 33 | 34
Completed | 29 | 29 | 32
Not Completed | 3 | 4 | 2
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal due to Caregiver Circumstances | 0 | 1 | 0
Not completed — Incorrectly Enrolled | 0 | 1 | 0
Period: Open-label Period (22 Weeks)
Arm/Group | 5 Milligram (mg) Tirzepatide/5 mg Tirzepatide | 10 mg Tirzepatide/10 mg Tirzepatide | Placebo/5 mg Tirzepatide
Started (A total of 90 participants continued study treatment at open label period. However, as per safety analysis set 2 overall N = 97 participants had atleast one dose of tirzepatide which was used for overall study safety assessments.) | 29 | 29 | 32
Safety Analysis Set 2 (Safety Analysis set 2 is defined as data obtained from mITT participants (those who took at least 1 dose of Tirzepatide was included in the analyses) during the double-blind period, open-label period, and safety follow-up period, regardless of adherence to study intervention or initiation of rescue antihyperglycemic medication.) | 32 | 33 | 32
Completed | 29 | 29 | 32
Not Completed | 0 | 0 | 0
Period: Safety Follow-up Period (4 Weeks)
Arm/Group | 5 Milligram (mg) Tirzepatide/5 mg Tirzepatide | 10 mg Tirzepatide/10 mg Tirzepatide | Placebo/5 mg Tirzepatide
Started | 29 | 29 | 32
Completed | 29 | 29 | 32
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 5 mg Tirzepatide: Participants received 5 mg Tirzepatide QW administered as SC injection via SDP for 30 weeks in double-blind period.
- 10 mg Tirzepatide: Participants received 10 mg Tirzepatide QW administered as SC injection via SDP for 30 weeks in double-blind period.
- Placebo: Participants received placebo QW administered as SC injection via SDP for 30 weeks in double-blind period.
- Total: Total of all reporting groups
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | Placebo | Total
Number analyzed (Participants) | 32 | 33 | 34 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.00 (1.93) | 14.60 (1.83) | 14.60 (1.79) | 14.70 (1.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 21 | 60
  Male | 11 | 15 | 13 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 17 | 24 | 65
  Not Hispanic or Latino | 8 | 16 | 9 | 33
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 5 | 8 | 20
  Asian | 1 | 2 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 0 | 3
  Black or African American | 5 | 4 | 2 | 11
  White | 17 | 19 | 21 | 57
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 1 | 1 | 0 | 2
  Brazil | 8 | 5 | 3 | 16
  India | 1 | 2 | 3 | 6
  Israel | 1 | 4 | 3 | 8
  Italy | 0 | 2 | 1 | 3
  Mexico | 10 | 8 | 13 | 31
  United Kingdom | 0 | 0 | 1 | 1
  United States | 11 | 11 | 10 | 32
Hemoglobin A1c [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time.
  Percentage of HbA1c | 8.22 (1.17) | 7.89 (1.22) | 8.02 (1.30) | 8.04 (1.23)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) (Pooled Doses of Tirzepatide 5 mg and 10 mg)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. Least Squares (LS) mean was determined by ANCOVA model for endpoint measures: Variable = Baseline + Baseline Antihyperglycemic medication + Baseline Age group + Treatment (Type III sum of squares)
Time Frame: Baseline, Week 30
Population: All randomized participants who received at least one dose of study drug and had evaluable data for this outcome obtained during the double-blind period regardless of adherence to study intervention or initiation of rescue antihyperglycemic medication.This analysis was planned to measure the outcome by combining the 5 mg tirzepatide treatment arm and 10 mg tirzepatide treatment arm as pooled doses of tirzepatide (5 mg/10 mg).
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Groups:
- Pooled Doses of Tirzepatide (5 mg, 10 mg): Participants received either 5 mg or 10 mg Tirzepatide QW administered as SC injection via SDP for 30 weeks in double-blind period.
Arm/Group | Pooled Doses of Tirzepatide (5 mg, 10 mg) | Placebo
Number analyzed (Participants) | 56 | 32
percentage of HbA1c | -2.03 (0.165) | -0.23 (0.229)
Statistical Analysis 1: Comparison: Pooled Doses of Tirzepatide (5 mg, 10 mg) vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean difference (Final Values) = -1.80, 95% CI 2-sided [-2.35 to -1.25]

2. Secondary Outcome: Change From Baseline in HbA1c (Individual Doses)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. LS mean was determined by ANCOVA model for endpoint measures: Variable = Baseline + Baseline Antihyperglycemic medication + Baseline Age group + Treatment (Type III sum of squares).
Time Frame: Baseline, Week 30
Population: All randomized participants who received at least one dose of study drug and had evaluable data for this outcome obtained during the double-blind period regardless of adherence to study intervention or initiation of rescue antihyperglycemic medication.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | Placebo
Number analyzed (Participants) | 29 | 27 | 32
percentage of HbA1c | -1.90 (0.236) | -2.16 (0.232) | -0.23 (0.229)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean difference (Final Values) = -1.67, 95% CI 2-sided [-2.31 to -1.02]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean difference (Final Values) = -1.93, 95% CI 2-sided [-2.57 to -1.29]

3. Secondary Outcome: Percentage of Participants Who Achieve ≤6.5% of HbA1c
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. Imputed data includes observed value and imputed value if endpoint measure is missing.
Time Frame: Week 30
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Groups:
- Pooled Doses of Tirzepatide (5mg,10mg): Participants received either 5 mg or 10 mg Tirzepatide QW administered as SC injection via SDP for 30 weeks in double-blind period.
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | Pooled Doses of Tirzepatide (5mg,10mg) | Placebo
Number analyzed (Participants) | 32 | 33 | 65 | 34
percentage of participants | 66.4 | 80.6 | 73.6 | 28.2
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 40.1, 95% CI 2-sided [18.6 to 61.7]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 51.6, 95% CI 2-sided [31.1 to 72.2]
Statistical Analysis 3: Comparison: Pooled Doses of Tirzepatide (5mg,10mg) vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 45.8, 95% CI 2-sided [27.5 to 64.1]

4. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) Standard Deviation Score (Age and Sex-matched)
Description: BMI SDS (age and sex matched), calculated using the World Health Organization (WHO) growth reference standards. BMI is calculated as weight in kilograms divided by height in meters squared (kg/m²) and converted to a Z-score (SDS) based on WHO reference data. A Z-score of 0 represents the population mean for a given age and sex. A BMI SDS between -1 and +1 is considered normal. Obesity is defined as BMI SDS > +2. Reductions in BMI SDS indicate improvement in weight status for individuals with obesity.
  LS mean was determined by the ANCOVA model for endpoint measures: Variable = Baseline + Baseline Antihyperglycemic medication + Baseline Age group + Treatment (Type III sum of squares)
Time Frame: Baseline, Week 30
Population: All randomized participants who received at least one dose of study drug and had evaluable data for this outcome obtained during the double-blind period regardless of adherence to the study intervention or initiation of rescue antihyperglycemic medication.
Measure: Least Squares Mean (Standard Error); unit: Z-score
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | Pooled Doses of Tirzepatide (5mg,10mg) | Placebo
Number analyzed (Participants) | 29 | 29 | 58 | 34
Z-score | -0.45 (0.072) | -0.76 (0.072) | -0.60 (0.050) | -0.09 (0.069)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean difference (Final Values) = -0.36, 95% CI 2-sided [-0.55 to -0.16]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean difference (Final Values) = -0.66, 95% CI 2-sided [-0.86 to -0.47]
Statistical Analysis 3: Comparison: Pooled Doses of Tirzepatide (5mg,10mg) vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean difference (Final Values) = -0.51, 95% CI 2-sided [-0.68 to -0.34]

5. Secondary Outcome: Change From Baseline in Fasting Serum Glucose (FSG)
Description: LS mean was determined by ANCOVA model for endpoint measures: Variable = Baseline + Baseline Antihyperglycemic medication + Baseline Age group + Treatment (Type III sum of squares).
Time Frame: Baseline, Week 30
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: milligram per deciliter (mg/dL)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | Pooled Doses of Tirzepatide (5mg,10mg) | Placebo
Number analyzed (Participants) | 28 | 28 | 56 | 33
milligram per deciliter (mg/dL) | -35.5 (7.76) | -50.6 (7.40) | -43.0 (5.42) | -6.6 (7.36)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p = 0.007, ANCOVA; LS Mean difference (Final Values) = -28.9, 95% CI 2-sided [-49.7 to -8.0]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean difference (Final Values) = -44.0, 95% CI 2-sided [-64.3 to -23.6]
Statistical Analysis 3: Comparison: Pooled Doses of Tirzepatide (5mg,10mg) vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean difference (Final Values) = -36.4, 95% CI 2-sided [-54.2 to -18.6]

6. Secondary Outcome: Percent Change From Baseline in BMI
Description: as for outcome 5
Time Frame: Baseline, Week 30
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent Change of BMI
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | Pooled Doses of Tirzepatide (5mg,10mg) | Placebo
Number analyzed (Participants) | 29 | 29 | 58 | 34
Percent Change of BMI | -6.73 (1.155) | -11.07 (1.154) | -8.90 (0.808) | -0.55 (1.107)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean difference (Final Values) = -6.18, 95% CI 2-sided [-9.31 to -3.05]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean difference (Final Values) = -10.52, 95% CI 2-sided [-13.67 to -7.38]
Statistical Analysis 3: Comparison: Pooled Doses of Tirzepatide (5mg,10mg) vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean difference (Final Values) = -8.35, 95% CI 2-sided [-11.05 to -5.66]

7. Secondary Outcome: Percentage of Participants Who Achieve <5.7% of HbA1c
Description: as for outcome 3
Time Frame: Week 30
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | Pooled Doses of Tirzepatide (5mg,10mg) | Placebo
Number analyzed (Participants) | 32 | 33 | 65 | 34
percentage of participants | 44.1 | 56.2 | 50.2 | 15.9
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p = 0.006, Regression, Logistic; Risk Difference (RD) = 29.5, 95% CI 2-sided [8.6 to 50.3]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 39.5, 95% CI 2-sided [18.8 to 60.2]
Statistical Analysis 3: Comparison: Pooled Doses of Tirzepatide (5mg,10mg) vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 34.6, 95% CI 2-sided [17 to 52.1]

8. Secondary Outcome: Percentage of Participants Who Achieve <7.0% of HbA1c
Description: as for outcome 3
Time Frame: Week 30
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | Pooled Doses of Tirzepatide (5mg,10mg) | Placebo
Number analyzed (Participants) | 32 | 33 | 65 | 34
percentage of participants | 79.6 | 84.5 | 82.1 | 37.4
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 43.4, 95% CI 2-sided [22.3 to 64.4]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 47.1, 95% CI 2-sided [26.4 to 67.7]
Statistical Analysis 3: Comparison: Pooled Doses of Tirzepatide (5mg,10mg) vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 45.2, 95% CI 2-sided [26.3 to 64.1]

9. Secondary Outcome: Percent Change From Baseline for Serum Lipid Levels
Description: Geometric LS mean was determined by the MMRM model for post-baseline measures: log(Actual Measurement/Baseline) = log(Baseline) + Baseline Antihyperglycemic medication + Baseline Age group + Treatment + Time + Treatment*Time (Type III sum of squares). Variance-Covariance structure (Change from Baseline) = Unstructured.
Time Frame: Baseline, Week 30
Population: as for outcome 2
Measure: Geometric Least Squares Mean (Standard Error); unit: Percent change of Serum Lipid Levels
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | Pooled Doses of Tirzepatide (5mg,10mg) | Placebo
Number analyzed (Participants) | 27 | 28 | 55 | 32
Percent change of Serum Lipid Levels
  Serum Cholesterol | -8.07 (2.319) | -13.82 (2.115) | -10.99 (1.564) | 5.07 (2.456)
  Serum High-density lipoprotein (HDL) Cholesterol 3RD generation, enzymatic | 5.56 (3.269) | 1.72 (3.087) | 3.62 (2.247) | 0.92 (2.887)
  Serum Triglycerides | -27.6 (4.816) | -35.8 (4.165) | -31.8 (3.165) | -1.74 (6.022)
  Serum low-density lipoprotein (LDL) Cholesterol Combined | -6.08 (3.870) | -11.97 (3.540) | -9.07 (2.618) | 9.84 (4.185)
  Serum very low-density lipoprotein (VLDL) Cholesterol Combined | -25.9 (5.005) | -34.8 (4.293) | -30.5 (3.276) | -0.26 (6.211)

10. Secondary Outcome: Change From Baseline in Height Standard Deviation Score (SDS)
Description: Height SDS (age and sex-matched), calculated using the World Health Organization (WHO) growth reference standards. Height SDS is derived by comparing a child's height to the median height for their age and sex in the WHO reference population, then expressing the difference in standard deviation units (Z-scores). A Z-score of 0 represents the population mean. A Height SDS below -2 indicates short stature. Positive changes in Height SDS from baseline reflect improvement in growth velocity or catch-up growth.
  LS mean was determined by MMRM model for post-baseline measures: Variable = Baseline + Baseline Age group + Baseline Antihyperglycemic medication + Treatment + Time + Treatment*Time(Type III sum of squares). Variance-Covariance structure (Actual Value) = Unstructured. Variance-Covariance structure (Change from Baseline) = Unstructured
Time Frame: Baseline, Week 30
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Z-score
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | Pooled Doses of Tirzepatide (5mg,10mg) | Placebo
Number analyzed (Participants) | 29 | 29 | 58 | 34
Z-score | -0.092 (0.0275) | -0.11 (0.0274) | -0.100 (0.0194) | -0.11 (0.0259)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p = 0.708, Mixed Models Analysis; LS Mean difference (Final Values) = 0.014, 95% CI 2-sided [-0.061 to 0.089]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p = 0.976, Mixed Models Analysis; LS Mean difference (Final Values) = -0.001, 95% CI 2-sided [-0.076 to 0.074]
Statistical Analysis 3: Comparison: Pooled Doses of Tirzepatide (5mg,10mg) vs Placebo; Test type: Superiority; p = 0.841, Mixed Models Analysis; LS Mean difference (Final Values) = 0.007, 95% CI 2-sided [-0.058 to 0.071]

11. Secondary Outcome: Change From Baseline in Weight SDS
Description: Weight SDS, calculated using Centers for Disease Control and Prevention (CDC) growth reference standards. Weight SDS is derived by comparing a child's weight to median weight for their age and sex in the CDC reference population, then expressing the difference in standard deviation units (Z-scores). A Z-score of 0 represents the population mean for a given age and sex. A Weight SDS below -2 may indicate underweight status, while a Weight SDS above +2 may indicate overweight or obesity. Change from baseline Weight SDS reflects shifts in growth trajectory, with positive changes indicating weight gain and negative changes indicating weight reduction.
  LS mean was determined by MMRM model for post-baseline measures: Variable = Baseline + Baseline Age group + Baseline Antihyperglycemic medication + Treatment + Time + Treatment*Time(Type III sum of squares). Variance-Covariance structure (Actual Value) = Unstructured. Variance-Covariance structure (Change from Baseline) = Unstructured
Time Frame: Baseline, Week 30
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Z-score
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | Pooled Doses of Tirzepatide (5mg,10mg) | Placebo
Number analyzed (Participants) | 29 | 29 | 58 | 34
Z-score | -0.38 (0.0600) | -0.50 (0.0594) | -0.44 (0.0422) | -0.099 (0.0570)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -0.29, 95% CI 2-sided [-0.45 to -0.12]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -0.4, 95% CI 2-sided [-0.57 to -0.24]
Statistical Analysis 3: Comparison: Pooled Doses of Tirzepatide (5mg,10mg) vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -0.34, 95% CI 2-sided [-0.49 to -0.2]

12. Secondary Outcome: Change From Baseline in Pediatric Quality of Life Inventory (PedsQL) Generic Core Scale
Description: The PedsQL Measurement Model measures health-related quality of life (HRQOL) in children (ages 8 to 12) and teenagers (ages 13 to 18). The 23-item PedsQL Generic Core Scale includes physical, emotional, social, and school functioning dimensions. The PedsQL Generic Core yields two summary scores: Physical Summary and Psychosocial Summary. Scores are transformed on a 0-100 scale, with higher scores indicating better functioning. Each item is scored from 0 (never) to 4 (almost always). Items are reverse scored and linearly transformed to a 0-100 scale so that higher scores indicate better HRQOL; the total score therefore ranges from 0 (worst) to 100 (best). Higher scores indicate better health-related quality of life. LS mean was determined by the MMRM model for post-baseline measures: Variable = Baseline + Baseline Antihyperglycemic Medication + Baseline Age Group + Treatment + Time + Treatment*Time (Type III sum of squares). Variance-Covariance structure (Actual Value) = Unstructured.
Time Frame: Baseline, Week 52
Population: All randomized participants who received at least one dose of study drug and had evaluable data for this outcome obtained during the double-blind, open-label, and safety follow-up periods regardless of adherence to study intervention or initiation of rescue antihyperglycemic medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- 5 mg Tirzepatide: Participants received 5 mg Tirzepatide once weekly (QW) administered as subcutaneous (SC) injection via single-dose pen (SDP) for 30 weeks in double-blind period and 22 weeks in open-label period
- 10 mg Tirzepatide: Participants received 10 mg Tirzepatide QW administered as SC injection via SDP for 30 weeks in double-blind period and 22 weeks in open-label period
- Placebo/5 mg Tirzepatide: Participants who received placebo QW administered as SC injection via SDP for 30 weeks in double-blind period were administered with 5 mg Tirzepatide QW administered as SC injection via SDP for 22 weeks in open-label period.
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | Placebo/5 mg Tirzepatide | Pooled Doses of Tirzepatide (5mg,10mg)
Number analyzed (Participants) | 29 | 27 | 25 | 56
score on a scale
  Physical Functioning Score | 4.26 (2.034) | 3.06 (2.092) | 5.03 (2.142) | 3.66 (1.456)
  Emotional Functioning Score | 4.35 (3.506) | 4.11 (3.601) | 6.78 (3.705) | 4.23 (2.514)
  Social Functioning Score | 4.16 (2.628) | 3.00 (2.696) | 4.54 (2.764) | 3.58 (1.878)
  School Functioning Score | 13.30 (3.095) | 0.18 (3.152) | 12.03 (3.239) | 6.74 (2.197)
  Psychosocial Health Summary Score | 7.82 (2.482) | 2.20 (2.533) | 7.47 (2.605) | 5.01 (1.767)
  Physical Health Summary Score | 4.26 (2.034) | 3.06 (2.092) | 5.03 (2.142) | 3.66 (1.456)
  Total Score | 6.65 (2.114) | 2.45 (2.163) | 6.61 (2.220) | 4.55 (1.507)

13. Secondary Outcome: Change From Baseline PedsQL (3.2) Diabetic Module
Description: The PedsQL 3.2 Diabetes Module has 33 items for ages 13 years and older, and 32 items (1 less item for the Worry Scale) for ages 2 to 12 years. The 5 dimensions consist of diabetes symptoms (15 items), treatment barriers (5 items), treatment adherence (6 items), worry [2 items (3 for teens and adults)] and communication (4 items). Item scaling is a 5-point scale from 0 (never) to 4 (almost always). Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. Higher scores reflect fewer problems and better functioning. LS mean was determined by MMRM model for post-baseline measures: Variable = Baseline + Baseline Antihyperglycemic medication + Baseline Age group + Treatment + Time + Treatment*Time(Type III sum of squares). Variance-Covariance structure (Actual Value) = Unstructured. Variance- Covariance structure (Change from Baseline) = Unstructured.
Time Frame: Baseline, Week 52
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | Placebo/5 mg Tirzepatide | Pooled Doses of Tirzepatide (5mg,10mg)
Number analyzed (Participants) | 29 | 27 | 25 | 56
score on a scale
  Diabetes Management Summary Score | 7.21 (2.669) | 8.60 (2.733) | 5.25 (2.872) | 7.90 (1.907)
  Total Score | 8.79 (2.310) | 8.74 (2.374) | 6.03 (2.489) | 8.76 (1.657)

14. Secondary Outcome: Population Pharmacokinetics (PopPK): Steady State Area Under the Concentration Curve (AUC) of Tirzepatide
Description: The steady-state AUCs were estimated from Tirzepatide concentrations at Weeks 0, 7, 16, and 29 using the population PK model by treatment group.
Time Frame: Week 0: after the first dose anytime on the same day. Weeks 7, 16, and 29: 1 to 24 hours, 24 to 96 hours, or 120 to 168 hours post-dose, as assigned by IWRS.
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data obtained during the double-blind period regardless of adherence to study intervention or initiation of rescue antihyperglycemic medication.
Measure: Mean (95% Confidence Interval); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide
Number analyzed (Participants) | 32 | 31
nanogram*hour per milliliter (ng*hr/mL) | 92100 [85700 to 98600] | 184000 [171000 to 197000]

ADVERSE EVENTS:
Time Frame: Baseline Up to Week 56
Description: All randomised participants who received at least one dose of study drug were included in safety analyses, regardless of adherence or use of rescue medication. Gender-specific events reflect adjusted at-risk counts.
  Per analysis plan, adverse events were reported for all mITT participants by randomized arms; for the double-blind period using safety analysis set 1; and for overall study using Safety Analysis Set 2, with combined data from Double blind, Open-Label and Safety Follow-Up Periods.
Groups:
- 5 mg Tirzepatide / Double-Blind Period: Participants received 5 mg of tirzepatide QW administered as SC injection via SDP for 30 weeks in a double-blind period.
- TZP 10mg / Double-Blind Period: Participants received 10 mg of tirzepatide QW administered as SC injection via SDP for 30 weeks in a double-blind period.
- Placebo / Double-Blind Period: Participants received placebo QW administered as SC injection via SDP for 30 weeks in a double-blind period.
- TZP 5mg / 5mg Open-Label and Safety Follow-Up Period: Participants who received 5 mg tirzepatide during the double-blind period continued to receive 5 mg of tirzepatide QW administered as SC injection via SDP for 22 weeks in the open-label period and 4 weeks in the safety follow-up period.
- TZP 10mg / 10mg Open-Label and Safety Follow-Up Period: Participants who received 10 mg of tirzepatide during the double-blind period continued to receive 10 mg of tirzepatide QW administered as SC injection via SDP for 22 weeks in the open-label period and 4 weeks in the safety follow-up period.
- Placebo/TZP 5mg Open-Label and Safety Follow-Up Period: Participants who received placebo QW during the double-blind period were switched to 5 mg tirzepatide QW administered as SC injection via SDP for 22 weeks in the open-label period and 4 weeks in the safety follow-up period.
Arm/Group | 5 mg Tirzepatide / Double-Blind Period | TZP 10mg / Double-Blind Period | Placebo / Double-Blind Period | TZP 5mg / 5mg Open-Label and Safety Follow-Up Period | TZP 10mg / 10mg Open-Label and Safety Follow-Up Period | Placebo/TZP 5mg Open-Label and Safety Follow-Up Period
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/33 | 0/34 | 0/32 | 0/33 | 0/32
Serious Adverse Events (participants affected / at risk) | 1/32 | 1/33 | 1/34 | 1/32 | 1/33 | 0/32
Other Adverse Events (participants affected / at risk) | 17/32 | 19/33 | 11/34 | 10/32 | 7/33 | 8/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Tirzepatide / Double-Blind Period (N=32) | TZP 10mg / Double-Blind Period (N=33) | Placebo / Double-Blind Period (N=34) | TZP 5mg / 5mg Open-Label and Safety Follow-Up Period (N=32) | TZP 10mg / 10mg Open-Label and Safety Follow-Up Period (N=33) | Placebo/TZP 5mg Open-Label and Safety Follow-Up Period (N=32)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Borderline personality disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 5 mg Tirzepatide / Double-Blind Period (N=32) | TZP 10mg / Double-Blind Period (N=33) | Placebo / Double-Blind Period (N=34) | TZP 5mg / 5mg Open-Label and Safety Follow-Up Period (N=32) | TZP 10mg / 10mg Open-Label and Safety Follow-Up Period (N=33) | Placebo/TZP 5mg Open-Label and Safety Follow-Up Period (N=32)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (18) | 4 (4) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 8 (23) | 8 (11) | 2 (7) | 5 (6) | 1 (1) | 6 (13)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (27) | 6 (7) | 3 (3) | 2 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (7) | 4 (24) | 1 (1) | 1 (1) | 2 (2) | 1 (3)
Injection site reaction (General disorders) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (3) | 2 (3) | 3 (3) | 1 (1)
Tonsillitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (7) | 3 (5) | 1 (1) | 3 (4) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 2 (3) | 2 (2) | 1 (3) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/21 (0) | 0/18 (0) | 0/21 (0) | 2/21 (8) | 0/18 (0) | 0/20 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT05260021/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-15): https://cdn.clinicaltrials.gov/large-docs/21/NCT05260021/SAP_001.pdf